CLINICAL TRIAL: NCT03457649
Title: A Phase I, Randomized, Double-Blind, Placebo-Controlled, SAD and MAD Intravenous Dose Study to Assess the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Immunogenicity of ARGX-113 in Healthy Males and Female Subjects
Brief Title: IV Dose Study to Assess the Safety, Tolerability, PK, PD and Immunogenicity of ARGX-113 in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: ARGX-113-1501
Record Dates: First submitted 2018-02-09; First posted 2018-03-07 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2018-02

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — efgartigimod alfa

STUDY DESIGN:
Intervention Model Description: SAD MAD
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ARGX-113 (Active Comparator): SAD and MAD with test product at different increasing doses
  Interventions: Biological: ARGX-113
- Placebo (Placebo Comparator): SAD and MAD with placebo at different increasing doses
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: ARGX-113
  Arms: ARGX-113
Biological: Placebo
  Arms: Placebo

SUMMARY:
A phase 1 study in healthy volunteers (female and male) to evaluate through SAD and MAD, the safety, PK, PD and immunogenicity of ARGX-113 administered intravenously.

DETAILED DESCRIPTION:
The phase 1 in healthy volunteers include:

SAD with 5 doses of test product and placebo

MAD with 2 doses and two dosing intervals of the test product and placebo

The safety, pharmacokinetics, pharmacodynamics and immunogenicity of the test product are evaluated.

ELIGIBILITY:
Inclusion Criteria:

Subjects meeting all of the following criteria are eligible to participate in this study:

1. Willingness and ability to understand the purpose and risks of the study and provide signed and dated informed consent prior to any procedures and be available for all study visits.
2. Male or female of non-child bearing potential, between 18-55 years of age, inclusive, on the day of signing the Informed Consent Form (ICF).
3. Body mass index (BMI) between 18-30 kg/m2, inclusive with a weight of at least 50 kg and no more than 100 kg.
4. Female subjects must have a negative blood pregnancy test at screening and a negative urine pregnancy test at Day -1.
5. Female subjects who are postmenopausal or surgically sterile (having had a hysterectomy, bilateral oophorectomy, or tubal ligation). Determination of serum follicle-stimulating hormone (FSH) will be done with FSH levels > 35 mIU/mL being confirmative for menopause. For hysterectomy and tubal ligation, documented confirmation will be requested.
6. Non-vasectomized male subjects having a female partner of childbearing potential must agree to the use of an effective method of contraception until 90 days after the last administration of study drug.
7. Male subjects have to agree not to donate sperm until 90 days after the last administration of study drug.
8. Judged by the investigator to be in good health based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and laboratory findings.
9. Discontinuation of all medications (including over-the-counter and/or prescription medication, dietary supplements, neutraceuticals, vitamins and/or herbal supplements such as Ginkgo biloba or Saint John's wort), except occasional paracetamol use (maximum dose of 2 g/day and maximum of 10 g/2 weeks), at least 2 weeks prior to the first study drug administration. In addition, subjects must agree to the prohibitions and restrictions for this study.
10. Non-smokers, and not using any nicotine-containing products. A non-smoker is defined as an individual who has abstained from smoking for at least 1 year prior to the screening.
11. Negative urine drug screen (amphetamines, barbiturates, benzodiazepines, cannabis, cocaine, opiates, methadone, and tricyclic antidepressants) at screening and Day -1.
12. Negative alcohol breath test at screening and Day-1. Note: A retest can be done in case of an out of range clinical laboratory test value that will determine a subject's eligibility. This retest should preferably be done at an unscheduled visit. The result of the retest will be considered for subject eligibility. If the retest is outside normal reference ranges, the subject may be included only if the investigator judges the abnormalities to be not clinically significant.

Exclusion Criteria:

Subjects meeting any of the following criteria are excluded from participation in this study:

1. Known hypersensitivity to study drug ingredients or a significant allergic reaction to any drug as determined by the investigator, such as anaphylaxis requiring hospitalization.
2. Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or any history of hepatitis from any cause with the exception of hepatitis A.
3. History of or a current immunosuppressive condition (e.g., human immunodeficiency virus [HIV] infection).
4. History of or evidence of active or latent or inadequately treated infection with Mycobacterium tuberculosis (TB) diagnosed by a positive QuantiFERON® TB-Gold In Tube test or a positive tuberculin skin test ("Mantoux") in case of a weak positive QuantiFERON® TB-Gold In Tube test.
5. Subjects with known clinically relevant immunological disorders.
6. History of severe allergic or anaphylactic reactions.
7. Symptoms of clinically significant illness in the 3 months before the initial study drug administration.
8. Presence or having sequelae of gastrointestinal, liver, kidney or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
9. History of malignancy within the past 5 years (except for basal cell carcinoma of the skin that has been treated with no evidence of recurrence).
10. Clinically relevant abnormalities detected on ECG regarding either rhythm or conduction (e.g., QTcF > 450 ms [male subjects] or >470 [female subjects], or a known long QT syndrome). A first degree heart block or sinus arrhythmia will not be considered as a significant abnormality.
11. Clinically relevant abnormalities detected on vital signs
12. Significant blood loss (including blood donation [> 500 mL]), or had a transfusion of any blood product within 12 weeks prior to the initial study drug administration or plan one within 4 weeks after the end of the study.
13. Treatment with any drug known to have a well-defined potential for toxicity to a major organ in the last 3 months preceding the initial study drug administration.
14. The subject has a history of consuming more than 21 (14 for females) units of alcoholic beverages per week or has a history of alcoholism or drug/chemical/substance abuse within past 2 years prior to screening (Note: one unit = 330 mL of beer, 110 mL of wine or 28 mL of spirits). Consumption of a large quantity of coffee, tea (> 6 cups per day) or equivalent.
15. Administration of an injectable drug within 30 days prior to the initial study drug administration.
16. Concurrent participation, or participation within 8 weeks prior to the initial study drug administration in a drug/device or biologic investigational research study, or participation within 15 weeks prior to initial study drug administration in an investigational research study with biologic response modifier administration.
17. Administration of a vaccine within 60 days prior to initial study drug administration.
18. Administration of any systemic immunosuppressant agent within 6 months prior to initial study drug administration.
19. Administration of any systemic steroid within 2 months prior to initial study drug administration;
20. Use of a prohibited therapy within 14 days prior to initial study drug administration.
21. Investigator or any sub-investigator, research assistant, pharmacist, study coordinator, or other staff or relative thereof who is directly involved in the conduct of the study.
22. Any condition or circumstances that in the opinion of the investigator may make a subject unlikely or unable to complete the study or comply with study procedures and requirements.
23. Pregnant or lactating women or women of childbearing potential.
24. Unsuitable vein for infusion and/or blood sampling.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 62 (Actual)
Dates: Start 2015-09-09 (Actual); Primary Completion 2016-11-15 (Actual); Study Completion 2017-02-21 (Actual)

PRIMARY OUTCOMES:
Number of (related) treatment emergent AE of single ascending dose of ARGX-113 | 57 days
  Determining the incidence, severity, and dose relationship of adverse events that are related to treatment with ARGX-113

SECONDARY OUTCOMES:
Number of (related) treatment emergent AE of multiple ascending doses of ARGX-113 | 78 days
  Determining the incidence, severity, and dose relationship of adverse events that are related to treatment with ARGX-113

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ulrichts P, Guglietta A, Dreier T, van Bragt T, Hanssens V, Hofman E, Vankerckhoven B, Verheesen P, Ongenae N, Lykhopiy V, Enriquez FJ, Cho J, Ober RJ, Ward ES, de Haard H, Leupin N. Neonatal Fc receptor antagonist efgartigimod safely and sustainably reduces IgGs in humans. J Clin Invest. 2018 Oct 1;128(10):4372-4386. doi: 10.1172/JCI97911. Epub 2018 Jul 24. PMID 30040076